CLINICAL TRIAL: NCT00598962
Title: Open, Noncomparative Trial of Multidrug Regimens Containing Azithromycin and Rifabutin Administered Three Times Per Week for the Treatment of M. Avium Complex (MAC) Lung Disease
Brief Title: Use of Azithromycin and Rifabutin Administered 3 Times Weekly for the Treatment of M. Avium Complex (MAC) Lung Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at Tyler (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Richard J. Wallace, Jr., M.D., Chairman Department of Microbiology, The University of Texas Health Science Center at Tyler
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 426
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Mycobacterium Avium Complex
Keywords: MAC
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection | interventions — Azithromycin; Rifabutin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- azithromycin and rifabutin/rifampin (Experimental): Azithromycin and rifabutin/rifampin administered three times weekly.
  Interventions: Drug: Azithromycin; Drug: Rifabutin/rifampin

INTERVENTIONS:
Drug: Azithromycin — Dosage dependent on clinical factors such as age, weight and patient-specific health status
  Other Names: Zithromax
Drug: Rifabutin/rifampin
  Other Names: mycobutin/

SUMMARY:
To determine the safety and efficacy of azithromycin, rifabutin and ethambutol given three times weekly in the treatment of lung infection with M. avium complex(MAC)

DETAILED DESCRIPTION:
Azithromycin given 3 times weekly along with rifampin/rifabutin and ethambutol for treatment of MAC

ELIGIBILITY:
Inclusion Criteria:

* Meet American Thoracic Society criteria for nontuberculous lung disease: two or more AFB smear positive, culture positive sputums or bronchoscopic samples and/or two or more AFB smear negative respiratory samples with moderate to heavy growth (2+-4+); abnormal CXR consistent with M. avium lung disease; abnormal CXR consistent with M. avium lung disease; absence of other lung pathogens (except for the coexistence of M. abscessus).
* Age 18 and older
* Pretreatment isolate of M. avium complex available for MIC determination
* Baseline laboratory and clinical testing for baseline CBC, Chemistry (including liver enzymes), hearing test, visual acuity and color discrimination
* Available for long term followup

Exclusion Criteria:

* History of macrolide or rifamycins allergy
* Laboratory evidence of mycobacterial resistance to azithromycin
* Children less than 18 years of age
* If a menstruating female, not pregnant and on adequate birth control
* HIV+ or at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 1994-12 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Clinical and microbiological outcomes such as clinical symptoms and laboratory cultures | 6 months
  neg cultures X3 ( sputum conversion)

SECONDARY OUTCOMES:
Microbiological cultures | 1yr
  neg culture 1 yr on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Wallace Jr., M.D., Principal Investigator — The University of Texas Health Science Center at Tyler
Locations (1):
- The University of Texas Health Science Center at Tyler, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: No